CLINICAL TRIAL: NCT03008018
Title: An Open Label Ascending Dose Study Evaluating the Safety/Tolerability, Pharmacokinetic and Pharmacodynamic Effects of KA2507 in Patients With Solid Tumours
Brief Title: Safety,Tolerability and MTD KA2507 (HDAC6 Inhibitor) in Patients With Solid Tumours
Acronym: HDAC6i
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Karus Therapeutics Limited (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KTP-003
Record Dates: First submitted 2016-12-21; First posted 2017-01-02 (Estimated); Last update posted 2020-08-19 (Actual); Status verified 2020-08

CONDITIONS: Solid Tumor, Adult

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- KA2507 (HDAC6 inhibitor) (Other): This is a single arm dose escalating study. Patients will be treated with open label KA2507 (HDAC6 inhibitor) capsules.
  Interventions: Drug: KA2507

INTERVENTIONS:
Drug: KA2507 — KA2507, an orally-active new chemical entity, is a potent and selective inhibitor of the HDAC6 enzyme, with potential clinical utility in the treatment of melanoma and other solid tumors. KA2507 has been shown to display potent in vitro activity in a range of cancer cell lines, including melanoma cell lines. KA2507 exerts potent in vivo efficacy in a syngeneic model of B16 melanoma. Here, the combination of the agent's direct tumor growth inhibition and metastasis suppression, coupled with its immunotherapeutic activity - demonstrated by decreased expression of STAT-3 and PD-L1 and increased expression of acetylated tubulin, gp100 and MHC Class I in tumors - have been observed.
  Other Names: HDAC6 Inhibitor; HDAC6i

SUMMARY:
The aim of the study is to evaluate the safety/tolerability, pharmacokinetic, and pharmaco-dynamic effects of KA2507 and establish the maximum tolerated dose (MTD). Patients with PD-L1 expressing solid tumors which have relapsed or are refractory to prior treatment will be eligible to participate in this study.

Following completion of the multiple ascending dose study, the protocol may be amended to include expansion cohorts in patients with melanoma and/or other solid tumors.

DETAILED DESCRIPTION:
The aim of the study is to evaluate the safety/tolerability, pharmacokinetic, and pharmaco-dynamic effects of KA2507 and establish the maximum tolerated dose (MTD). Patients with PD-L1 expressing solid tumors which have relapsed or are refractory to prior treatment will be eligible to participate in this study.

Following completion of the multiple ascending dose study, the protocol may be amended to include expansion cohorts in patients with melanoma and/or other solid tumors.

This is a multiple ascending dosing (MAD) study of up to 6 treatment regimens cohorts based on using a 3+3 design (up to 36 patients overall). The principal objective is to establish the maximum tolerated dose, safety, tolerability and pharmacokinetic (PK) profile in blood and urine of this HDAC6 inhibitor in patients with solid tumors and to explore effects on pharmacodynamic markers of target engagement and response to treatment.

Daily/twice daily doses will be given as open label monotherapy. A review of safety and PK data will be conducted once the last patient in each cohort reaches day 28 of treatment. The review will confirm the dose to be used for the subsequent cohort. Dose escalation will be continued until the MTD is reached. Upon completion of the dose escalation phase of the study, dose expansion phases will be planned.

Patients responding to treatment may elect to remain on therapy until disease progression, death or the investigator decides to stop treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years at the screening visit.
2. Patients with histologically or cytologically documented, confirmed diagnosis of advanced malignancy, whose disease failed to respond to or progressed after standard therapy or they could not tolerate standard therapy.
3. Measurable or evaluable disease according to RECIST v1.1.
4. ECOG performance status of 0 or 1.
5. Predicted life expectancy ≥12 weeks.
6. For men and women of child-bearing potential, willing to use adequate contraception (i.e., latex condom, cervical cap, diaphragm, abstinence, etc.) for the entire duration of the study.

1. If female, must be either postmenopausal, sterilised or, if sexually active, effectively practicing an acceptable method of contraception (either oral, parenteral, or implantable hormonal contraceptives, intrauterine device or barrier and spermicide). Subjects must agree to use adequate contraception during the study and for at least 12 weeks (or longer as per local requirement) after the last dose of study treatment.

2. Male subjects agree to ensure that they or their female partner(s) use adequate contraception during the study and for at least 12 weeks (or longer as per local requirement) after the subject receives their last dose of study treatment.

Exclusion Criteria:

1. Patients are not able to provide written informed consent to study participation
2. Patients who have been treated with most recent radiotherapy, hormonal therapy, immunotherapy, chemotherapy or investigational drugs within ≤21 days or 5 half-lives (whichever is shorter) from enrolment (screening), and/or who have any unresolved NCI Common Terminology Criteria of Adverse Events (CTCAE) v4.03 > Grade 1 treatment-related side effect (with the exception of alopecia).
3. Patient has anemia due to HbS or HbC disease, alpha or beta thalassaemia
4. Patient has Glucose-6-phosphate deficiency
5. Patient has known or suspected history of cytochrome b5-MetHb-reductase pathway deficiency
6. Persons of Navajo, Athabaska Alaskan or Siberian Yakutsk descent
7. Patient has untreated severe hypothyroidism
8. Patient has laboratory estimations indicating organ system dysfunction:

   1. Absolute neutrophil count (ANC) <1.5 X 109/L
   2. Platelets <100 X 109/L
   3. Hemoglobin <9g/dL
   4. Total bilirubin >1.5 mg/dL
   5. ALT and AST >3.0 times the ULN if no liver involvement or >5 times the ULN with liver involvement.
   6. Calculated creatinine clearance <60mL/min estimated using the Cockcroft-Gault equation:

      • Cockcroft-Gault equation: creatinine clearance = (140 - age in years) x (wt in kg)) x 1.23) / (serum creatinine in micromol/l) [For women multiply the result of calculation by 0.85].
9. Major surgery (excluding placement of vascular access) ≤21 days from beginning of the study drug or minor surgical procedures ≤7 days. No waiting is required following implantable port and catheter placement.
10. Any of the following cardiac criteria:

    1. Congestive heart failure (CHF), grade III or IV per New York Heart Association (NYHA) classification
    2. Symptomatic cardiomyopathy
    3. > Class II Cardiac ventricular arrhythmias requiring anti-arrhythmic therapy
    4. Unstable angina or new-onset angina
    5. QTcF interval >470 ms on screening ECG.

9. Severe or uncontrolled systemic diseases including uncontrolled hypertension, active bleeding diatheses 10. Any evidence of active infection including active Hepatitis B, Hepatitis C or human immunodeficiency virus 11. The patient has concurrent severe and/or uncontrolled medical disease that could compromise participation in the study (i.e., uncontrolled diabetes, severe infection requiring active treatment, severe malnutrition, chronic severe liver or renal disease, uncontrolled hypertension, active bleeding diatheses).

12. Active infection requiring IV antibiotics within two weeks prior to treatment, or evidence of TB infection.

13. Hepatitis B, Hepatitis C or human immunodeficiency virus 14. Previously untreated brain metastases. Patients who have received radiation or surgery for brain metastases are eligible if therapy was completed at least 3 weeks previously and there is no evidence of central nervous system disease progression, mild neurologic symptoms, and no requirement for chronic corticosteroid therapy.

15. Lactating, breastfeeding, or positive pregnancy test for female patients of child-bearing potential.

16. The patient is unable to swallow capsules and/or has a surgical or anatomical condition that precludes swallowing and absorbing oral medication on an ongoing basis (for oral therapy only).

17. Patients with prior stem cell transplantation or solid organ transplantation.

18. History of other malignancies (except for adequately treated basal or squamous cell carcinoma or carcinoma in situ) within the last 3 years.

17. Any other condition that would, in the investigator's judgment, contraindicate the patient's participation in the clinical study due to safety concerns or compliance with clinical study procedures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2017-08-07 (Actual); Primary Completion 2020-06-10 (Actual); Study Completion 2020-06-10 (Actual)

PRIMARY OUTCOMES:
The occurrence of dose limiting toxicity | 28 days
  1. Any event with possible or probable relationship to study drug occurring up to day 28 from the start of treatment as assessed using the National Cancers Institutes Common Terminology Criteria for Adverse events version 4.03 therapy.

SECONDARY OUTCOMES:
Concentration of KA2507 in plasma over time (hours) post dosing | 24 weeks
Concentration of KA2507 in urine over time (hours) post dosing | 24 weeks
Blood concentration of histone acetylation during KA2507 treatment | 24 weeks
Blood concentration of tubulin during KA2507 treatment | 24 weeks
Number of Participants With Abnormal Laboratory Values and/or Adverse Events That Are Related to Treatment | 24 weeks
Clinical outcomes using the RECIST 1.1 criteria | 24 weeks
Clinical outcomes using Immuno-RECIST criteria | 24 weeks

OTHER OUTCOMES:
Concentration of PD-L1 expression in tumor tissue | 24 weeks
Concentration of MHC-1 expression in tumor tissue | 24 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- M D Anderson, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Tsimberidou AM, Beer PA, Cartwright CA, Haymaker C, Vo HH, Kiany S, Cecil ARL, Dow J, Haque K, Silva FA, Coe L, Berryman H, Bone EA, Nogueras-Gonzalez GM, Vining D, McElwaine-Johnn H, Wistuba II. Preclinical Development and First-in-Human Study of KA2507, a Selective and Potent Inhibitor of Histone Deacetylase 6, for Patients with Refractory Solid Tumors. Clin Cancer Res. 2021 Jul 1;27(13):3584-3594. doi: 10.1158/1078-0432.CCR-21-0238. Epub 2021 May 4. PMID 33947698